CLINICAL TRIAL: NCT04636723
Title: Neuroinflammation in Chronic Systemic Symptoms (CSS): Proof-of-Concept Study Using PET and EEG/ERP Biomarkers
Brief Title: Neuroinflammation in Chronic Systemic Symptoms (CSS)
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Poppy Schoenberg, Principle Investigator, Vanderbilt University Medical Center
Other Study IDs: IRB #202009
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Cancer; Cancer Head Neck; Neuroinflammatory Response; Chronic Inflammation; Chronic Disease; Chronic Pain
Keywords: PET; EEG/ERP; MRI/DTI; Cytokine; Chemokine; Neurophysiology; Molecular Radiology
MeSH Terms: conditions — Neoplasms; Head and Neck Neoplasms; Chronic Disease; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HNC Patients w/ CSS: HNC survivor patients presenting high chronic systemic symptoms
- Healthy Controls: Non-clinical controls
- HNC Patients wo/ CSS: Patient Control - HNC survivor patients presenting no/low chronic systemic symptoms

SUMMARY:
The purpose of the present research protocol is to investigate and identify translocator protein 18kDa, MRI DTI, and EEG/ERPs, markers of Chronic Systemic Symptoms (CSS).

DETAILED DESCRIPTION:
In 2016, there were an estimated 15.5 million cancer survivors in the US, with a forecasted 20.3 million by 2026. Three percent of those survivors were treated for Head and neck cancers (HNC). This number is expected to rise due to increased long-term survival in patients with HPV associated oropharyngeal cancer. Increasing survivorship has generated a surge of interest in late effects of HNC therapy. Studies to date have largely focused on chronic effects stemming from local tissue damage. Recent data suggests that late systemic effects may be equally problematic. Chronic systemic symptoms (CSS) persist far longer than previously considered and are the source of significant function loss and detriment to quality of life. CSS include fatigue, neurocognitive dysfunction, centralized pain, mood disorders, sleep disturbances, and hypothalamic dysfunction manifested as thermal discomfort or hyperhidrosis. Systemic symptoms occur in clusters resulting in a heightened clinical impact. As with other critical illnesses, the trajectory of recovery from the systemic symptoms from cancer treatment is varied. Some patients will recover to baseline quickly post treatment while others display CSS that persist or worsen over time resulting in functional deficits, frailty, and an early aging phenotype which may impact survival. Survivors exhibiting a "slow burn" trajectory as manifested by persistent systemic symptom burden and worsening function over time, require extensive on-going long-term management. These patients often fail to return to work or previously held family roles. CSS may therefore be associated with greater economic cost than the initial treatment.

Work that spans a wide array of inflammatory disease processes (such as fibromyalgia, chronic fatigue syndrome, irritable bowel, etc.) demonstrate the presence of somatic, affective, and cognitive symptoms. Neuroinflammation is hypothesized to be the underlying cause of these symptoms and their manifestations. More specifically, peripheral injury/trauma/cancer release inflammatory mediators that activate glial components of peripheral and central cellular circuitry causing inflammation of the CNS. However, the concept that CSS is underlined by neuroinflammation is largely theoretical from disparate and indirect evidence. A gap in the evidence base suggests direct investigation of neuroinflammation in CSS patients in capturing a mechanistic marker is urgently needed in order to (1) present CSS as a diagnostic entity, (2) fully understand its neurobiological mechanism, and (3) test/develop appropriate treatments.

ELIGIBILITY:
* Inclusion Criteria for HNC patients:

  * Age ≥ 21
  * HNC of larynx, pharynx, oral cavity paranasal sinus, salivary gland, or unknown primary
  * Any histology of any epithelial origin
  * Completed therapy a minimum of 3 months prior to study entry
  * At least two systemic symptoms on the VHNSS-GSS subscale
  * Able to speak English to understand instructions and be able to provide informed consent
* Exclusion Criteria for HNC patients:

  * History of neurodegenerative disease, unrelated to cancer history/treatment
  * Alcohol/substance abuse/dependence within the last 6 months
  * Current or previous co-morbid bipolar disorder-, psychosis-, obsessive compulsive disorder-, eating disorders-, personality disorders-,
  * Neurological disorders unrelated to cancer and its treatment (e.g. ADHD, ASDs, epilepsy)
  * Learning difficulties.
* Inclusion Criteria for healthy controls:

  * Age ≥ 21
  * Able to speak English to understand instructions and be able to provide informed consent
* Exclusion Criteria for healthy controls:

  * History of HNC of larynx, pharynx, oral cavity paranasal sinus, salivary gland, or unknown primary
  * Alcohol/substance abuse/dependence within the last 6 months
  * Current or previous co-morbid bipolar disorder-, psychosis-, obsessive compulsive disorder-, eating disorders-, personality disorders-,
  * Neurological disorders (e.g. ADHD, ASDs, epilepsy)
  * Learning difficulties.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10x HNC patients will be recruited via Vanderbilt's Department of Otolaryngology.
  10x Healthy controls will be recruited via VUMC recruitment listserv and ResearchMatch.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Positron Emission Tomography (PET) | 12 months
  Centralized Microglial Activation measured via mitochondrial translocator protein 18kDa (TSPO).

SECONDARY OUTCOMES:
EEG/ERP concomitant to working memory neurobehavioral task | 12 months
  Cognitive function as recommended by the International Cognition and Cancer Task Force (ICCTF)
EEG/ERP concomitant to sustained attention neurobehavioral task | 12 months
  Cognitive function as recommended by the International Cognition and Cancer Task Force (ICCTF)
Diffusion Tensor Imaging (DTI) | 12 months
  Diffusion coefficients as measure of cellular inflammation
Peripheral Cytokine and Chemokine Inflammation | 12 months
  Blood marker Interleukin-6 (IL-6)
Peripheral Cytokine and Chemokine Inflammation | 12 months
  Blood marker C reactive protein (CRP)
Peripheral Cytokine and Chemokine Inflammation | 12 months
  Blood marker nuclear factor (NF)-kB transcription factor

OTHER OUTCOMES:
Clinical Measure: Vanderbilt Head and Neck Symptom Survey (VHNSS) version 2.0 plus general symptom survey (GSS) | 12 months
  Validated tool to measure physical symptom burden and functional deficits related to head/neck cancer and its treatment.
Clinical Measure: Neurotoxicity Rating Scale (NRS) | 12 months
  37 item tool examining neurocognitive symptoms associated with neurotoxicity of medical treatment.
Clinical Measure: Central Sensitivity Inventory (CSI) | 12 months
  Two-part survey consisting of 35 questions. Part A aims to identify frequency of experienced systemic symptoms. Part B determines previous diagnosis of Central Sensitivity Syndromes or related disorders.
Clinical Measure: Pain Inventory (PI) | 12 months
  Diagram in which patients document specific areas of pain in the body, and rate pain intensity on a scale 1-10 in the past 3 months (i.e. with scores 3+ constituting chronic pain).
Clinical Measure: Patient Reported Outcomes Measurement Information System (PROMIS-29) | 12 months
  assesses 7 domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, participation in social roles/activities) using 5-point Likert scale, across 29-items.
Clinical Measure: • Behavior Rating Inventory of Executive Function - Adult version (BRIEF-A) | 12 months
  Measures nine non-overlapping theoretically and empirically derived clinical domains: Inhibit, Self-Monitor, Plan/Organize, Shift, Initiate, Task Monitor, Emotional Control, Working Memory, and organization of Materials.

CONTACTS AND LOCATIONS:
Overall Officials: Poppy Schoenberg, PhD, Principal Investigator — Osher Center for Integrative Medicine, VANDERBILT UNIVERSITY MEDICAL CENTER
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will adhere to the NIH Sharing of Biomedical Research Resources: Guidelines for Recipients of NIH Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources.
  1. Quality-controlled raw data as well as processed data used in publications will be de-identified before sharing upon "reasonable request". As described in the proposal, workflows and structure will be exactly described in reports and documented to allow precisely reproduce results from raw data and replicate methodology. Final data (computerized datasets with raw data and derived variables) that have not yet been published will be shared in a timely manner.
  2. Software programs (i.e. experimental paradigm scripts produced for this study) and documentation will be made available for research purposes to replicate findings upon "reasonable request", and any software/script sharing requirements by journals.
Supporting Information: CSR
Time Frame: 24 months